CLINICAL TRIAL: NCT02305589
Title: The Comparison of Sugammadex and Conventional Cholinesterase Inhibitor on the Aspect of Postoperative Delirium in the Elderly Patients Undergoing Hip Surgery
Brief Title: The Clinical Changes Before and After Sugammadex in the Patients Undergoing Hip Surgery on the Aspect of Delirium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: KUH1160075
Record Dates: First submitted 2014-11-17; First posted 2014-12-02 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Delirium
Keywords: postoperative delirium; sugammadex; cholinesterase inhibitor; hip fracture surgery
MeSH Terms: conditions — Delirium; Emergence Delirium | interventions — Sugammadex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sugammadex — Muscle relax reversing agent
  Other Names: Bridion

SUMMARY:
This study evaluated the effect of sugammadex on postoperative delirium in elderly patients undergoing hip fracture surgery.

Medical records from 235 consecutive patients undergoing hip fracture surgery were retrospectively reviewed and total 61 patients were excluded for age under 60 years, preoperative neurologic problem. Finally total 174 patients aged over 60 years undergoing hip fracture surgery with general anaesthesia using a neuromuscular blocking agent from 2012 to 2014 at a university hospital were analyzed to compare perioperative incidence of postoperative delirium, pulmonary complications, intensive care unit (ICU) admission, and ICU and hospital stay duration and laboratory findings between patients treated with sugammadex (S group) and conventional cholinesterase inhibitors (C group).

DETAILED DESCRIPTION:
Study population The medical records of patients undergoing hip surgery under general anaesthesia with neuromuscular blocking agents at Konkuk University Medical Center from February 2012 to August 2014 review.

The patients were divided according to use (S group) or not (C group) of sugammadex for recovery from neuromuscular blocking agent.

exclusion criteria

1. age < 60 years
2. preoperative neurologic or psychological problem including dementia, Parkinson's disease or delirium
3. other concurrent surgery.

Assessment of postoperative delirium Evaluation of postoperative delirium was done in the general ward or in the ICU by the responsible surgeon using commonly accepted delirium symptoms in addition to the confusion assessment method (CAM) rating for delirium. Delirium symptoms were defined as the presence of any of the following: acute onset and fluctuating symptoms; inattention; speech disorganization; level of consciousness change; disorientation; memory impairment; perceptual disturbance; abnormal psychomotor activity; and altered sleep wake cycle. Incidence of postoperative delirium assess by medical records review.

Postoperative clinical follow-up

By medical records review, the following clinical data were obtained:

transfusion amount of packed red blood cell during intraoperative period and up to postoperative 24 hours postoperative visual analogue scale (VAS, ranging from 0 [no pain] to 100 [worst pain imaginable]) up to postoperative day 1; delayed extubation events up to postoperative day 7; postoperative pulmonary complication [new onset abnormal findings in postoperative chest radiography with pulmonary symptoms such as cough, sputum, dyspnea] up to postoperative day 7; postoperative hypoxia [oxygen saturation on pulse oximeter < 95%] up to postoperative 24 hours; the event of admission to ICU; duration of ICU stay; duration of hospital stay. Perioperative laboratory findings, Haemoglobin (Hb), haematocrit (Hct), and serum levels of total protein, albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatinine and high sensitivity C reactive protein (HS-CRP) during intraoperative period and up to postoperative 24 hours were assessed by medical records review.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing hip surgery under general anaesthesia with neuromuscular blocking agents

Exclusion Criteria:

1. age < 60 years
2. preoperative neurologic or psychological problem including dementia, Parkinson's disease or delirium
3. other concurrent surgery.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing hip surgery under general anaesthesia with neuromuscular blocking agents
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | up to postoperative 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D., Ph.D., Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Krenk L, Rasmussen LS. Postoperative delirium and postoperative cognitive dysfunction in the elderly - what are the differences? Minerva Anestesiol. 2011 Jul;77(7):742-9. PMID 21709661
- [Result] Zywiel MG, Prabhu A, Perruccio AV, Gandhi R. The influence of anesthesia and pain management on cognitive dysfunction after joint arthroplasty: a systematic review. Clin Orthop Relat Res. 2014 May;472(5):1453-66. doi: 10.1007/s11999-013-3363-2. PMID 24186470
- [Result] Plaud B, Debaene B, Donati F, Marty J. Residual paralysis after emergence from anesthesia. Anesthesiology. 2010 Apr;112(4):1013-22. doi: 10.1097/ALN.0b013e3181cded07. No abstract available. PMID 20234315